CLINICAL TRIAL: NCT03076177
Title: The Effectiveness of Kinesio Taping Method for Knee Osteoarthritis. Randomized Double Blinded Clinical Trial.
Brief Title: The Effectiveness of Kinesio Taping Method for Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: International Kinesio Taping association (Unknown)
Responsible Party: Principal Investigator, Venta Donec, Venta Donec, MD, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 1
Record Dates: First submitted 2016-09-12; First posted 2017-03-10 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis, kinesio taping, knee function, pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kinesio taping group (Experimental): Participants receiving kinesio taping application
  Interventions: Other: Taping application
- Non specific taping (Sham Comparator): Participants receiving non specific taping application
  Interventions: Other: Taping application

INTERVENTIONS:
Other: Taping application — Kinesio taping application will be applied for experimental group; non specific taping application for control
  Other Names: Kinesio taping/non specific taping

SUMMARY:
Purpose of our study is to evaluate effectiveness of Kinesio Taping method for knee osteoarthritis. Using simple concealed randomization procedure to form two groups (kinesio taping and control-nonspecific taping) of 100 knee osteoarthritis patients in each. 1 month all patients (depending on the group they will be allocated to) will receive either kinesio taping applications or non-specific taping: 4 applications per subject. Three times: before taping, after a month with tapes, and after 1 month without tapes evaluation of knee function, mobility, quality of life will be evaluated, including clinical examination of knee joint, measurements of knee flexion and extension by goniometer, circumference of leg over the knee, in ½ of thigh and in ½ of calf (to evaluate edema); pain will be evaluated by questionnaire, patella tendon algometry; force of calf flexors and extensors will be evaluated using Lovett manual muscle testing scale, goniometry for knee flexion/extension; for mobility, knee function, life quality evaluations - 10 Meter Walk , Five Times Sit to Stand Tests will be performed, Knee injury and Osteoarthritis Outcome Score (KOOS) and Medical Outcomes Study Short Form 36 2 version (SF-36 2v) questionnaires will be used. Also data about the need of analgesic medicament will be collected from subjects.

DETAILED DESCRIPTION:
After subject inclusion into research, two groups (study (kinesio taping) group and control-non specific taping) of 100 patients in each will be formed by the procedure of concealed randomization (person not connected with study by the help of random number generator will make allocation of subjects to the groups).

All subjects will receive taping (kinesio or non specific) for one month (tapes will be applied once a week, 4 times per person, held on skin for 6 days with one day break - without tape). Subjects will be allowed to use their conventional analgesic medicaments 'per os' or parenterally if needed. Control and Kinesio taping applications will be done by certified kinesio taping practitioner (CKTP) or other team member trained by CKTP (researcher 'B'). Other research team member (researcher 'A') will do evaluations of chosen criteria (pain, knee function, mobility etc.), he will not be informed to which group (kinesio taping or placebo) subject was allocated, the same researcher (researcher 'A') will do repeated evaluations for the same subject after first and second months of participation in study.

Taping applications:

Control. For non specific taping Kinesio Tape tex Gold finger print (FP) will be used, however tapes will be applied without using specific application manner of kinesio taping method. I.e. - tapes will be applied in subject lying position with knee fully extended using 0% of available tension 10 cm above and 10cm below superior and inferior poles of patella (approx 5x25cm) and on medial and lateral sides of knee joint (small pieces of tape approx. 5x5cm)

Kinesio taping. Kinesio Tape tex Gold FP will be used . Subjects will get two Y strips applied in lymphatic correction manner using paper off tension (tapes will be applied in fully flexed knee position); than two I strips will be applied for patella tendon and lateral and medial collateral ligaments using 75-100% of tension: over patella tendon - in fully flexed knee position, 100% of tension; over ligaments - in 20-30 degrees of knee flexion,75% of tension ; ends -with no tension, - seeking to increase stimulation of mechanoreceptors over the area, improve proprioception and reduce pain.

All subjects, before starting the research, will be informed in written as well as in spoken form about the research, it's type, goals, possible inconveniences (possible skin irritation, hair picking etc.). Every subject will have right to stop their participation in research at any time.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed (and radiologically verified) I-III stage knee osteoarthritis, has no contraindications (exclusion criteria) to participate in research, are willing to follow studies protocol and gives informed approval to participate in this research in written form.

Exclusion Criteria:

* Rheumatoid arthritis or other systemic rheumatoid disease (LE, sclerodermia,.. etc)
* Fragile, very sensitive skin or it's lesions in areas where tapes are to be applied
* Inability to do functional tests according study protocol due to very impaired knee function or severe comorbidities.
* Diagnosed or suspected cancer in areas where tapes to be applied
* < than 6 months after intra-articular injections in knee joint
* Constant usage of analgesic medicament due to comorbidities
* Pregnancy
* History of Kinesio Taping method applications in the past
* Need for orthotics
* Unwillingness not to use local ointments in knee region during participation in study period (i.e. 2 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2014-10; Primary Completion 2018-07 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Change in knee pain intensity from baseline at 4 weeks | 4 weeks
  Numeric Pain Rating Scale (an 11-point scale from 0-10. "0" = no pain, "10" = the most intense pain imaginable)

SECONDARY OUTCOMES:
Change in knee pain intensity from baseline at 8 weeks | 8 weeks
  Numeric Pain Rating Scale (an 11-point scale from 0-10. "0" = no pain, "10" = the most intense pain imaginable)
Change in patella tendon pain threshold from baseline at 4 weeks | 4 weeks
  measured with algometer (kgf)
Change in patella tendon pain threshold from baseline at 8 weeks | 8 weeks
  measured with algometer (kgf)
Change in knee function at 4 weeks from baseline | after 4weeks
  measured by KOOS which consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Change in knee function at 8 weeks from baseline | after 8 weeks
  measured by KOOS which consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Change in gait speed from baseline at 4 weeks | 4 weeks
  10 Meter Walk test (m/s)
Change in gait speed from baseline at 8 weeks | 8 weeks
  10 Meter Walk test (m/s)
Change in time needed for five times sit to stand test from baseline at 4 weeks | 4 weeks
  Five Times Sit to Stand Tests (s)
Change in time needed for five times sit to stand test from baseline at 8 weeks | 8 weeks
  Five Times Sit to Stand Tests (s)
Change in knee flexion from baseline at 4 weeks | 4 weeks
  measured active knee flexion in standardized position with goniometer (degrees)
Change in knee flexion from baseline at 8 weeks | 8 weeks
  measured active knee flexion in standardized position with goniometer (degrees)
Change in knee extension from baseline at 4 weeks | 4 weeks
  measured active knee extension in standardized position with goniometer (degrees)
Change in knee extension from baseline at 8 weeks | 8 weeks
  measured active knee extension in standardized position with goniometer (degrees)
Change in leg circumference (thigh, knee, calf) from baseline at 4 weeks | 4 weeks
  leg circumference with tape measured in standardized points of leg (thigh, knee, calf region) (cm)
Change in leg circumference (thigh, knee, calf) from baseline at 8 weeks | 8 weeks
  leg circumference with tape measured in standardized points of leg (thigh, knee, calf region) (cm)
Change in patient-reported outcome measure of health-related quality of life from baseline at 4 weeks | 4 weeks
  Medical Outcomes Study Short Form 36 2 version (SF-36v2) will be used. Measure is divided into 8 subscales and 2 composite domains
  The 8 subscales are:
  1. Physical Functioning
  2. Role Limitations due to Physical Problems
  3. General Health Perceptions
  4. Vitality
  5. Social Functioning
  6. Role Limitations due to Emotional Problems
  7. General Mental Health
  8. Health Transition Respondents are asked to answer items referring to the past 4 weeks Recommended scoring system for the SF-36 is a weighted Likert system for each item Items within subscales are totaled to provide a summed score for each subscale or dimension.
  Each of the 8 summed scores is linearly transformed onto a scale from 0 (negative health) to 100 (positive health) to provide a score for each subscale.
Change in patient-reported outcome measure of health-related quality of life from baseline at 8 weeks | 8 weeks
  Medical Outcomes Study Short Form 36 2 version (SF-36v2) will be used. Measure is divided into 8 subscales and 2 composite domains
  The 8 subscales are:
  1. Physical Functioning
  2. Role Limitations due to Physical Problems
  3. General Health Perceptions
  4. Vitality
  5. Social Functioning
  6. Role Limitations due to Emotional Problems
  7. General Mental Health
  8. Health Transition Respondents are asked to answer items referring to the past 4 weeks Recommended scoring system for the SF-36 is a weighted Likert system for each item Items within subscales are totaled to provide a summed score for each subscale or dimension.
  Each of the 8 summed scores is linearly transformed onto a scale from 0 (negative health) to 100 (positive health) to provide a score for each subscale.
Objective tolerance of taping (kinesio, non-specific) method | first 4 weeks of participation
  inspection of skin for any signs of redness, rash, etc., evaluated once every week
Subjective tolerance of taping (kinesio, non-specific) method | first 4 weeks of participation
  questionnaire for subjective evaluation of method from participants (side effects, inconveniences, skin problems, comments, opinion on pain relief and improvement on mobility) evaluated once every week
Change in need of analgesic medicament from baseline at 4 weeks | 4 weeks
  questionnaire about the need of analgesic medicament (type of drug, dose, frequency of use recorded)
Change in need of analgesic medicament from baseline at 8 weeks | 8 weeks
  questionnaire about the need of analgesic medicament (type of drug, dose, frequency of use recorded)

CONTACTS AND LOCATIONS:
Overall Officials: Raimondas Kubilius, PhD, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- LithuanianUHS, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Donec V, Kubilius R. The effectiveness of Kinesio Taping(R) for pain management in knee osteoarthritis: a randomized, double-blind, controlled clinical trial. Ther Adv Musculoskelet Dis. 2019 Aug 29;11:1759720X19869135. doi: 10.1177/1759720X19869135. eCollection 2019. PMID 31497072